CLINICAL TRIAL: NCT05376111
Title: A Prospective, Multi-Center Study to Evaluate the Efficacy and Safety of Venetoclax Combined With Azacitidine Regimen in Newly Diagnosed T-cell Acute Lymphoblastic Leukemia Patients
Brief Title: Study of Venetoclax Combined With Azacitidine Regimen in Newly Diagnosed T-ALL Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Northern Jiangsu People's Hospital (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZTALL01
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: T-cell Acute Lymphoblastic Leukemia; Recruiting
Keywords: Venetoclax; Azacitidine; T-ALL; Newly diagnosed
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetclax combined with Azacitidine (Experimental): T-cell acute lymphoblastic leukemia patients reveive venetoclax combined with azacitidine regimen treatment.
  Interventions: Drug: Venetoclax, Azacitidine

INTERVENTIONS:
Drug: Venetoclax, Azacitidine — Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-21); azacitidine 75 mg/m2 subcutaneously once daily on days 1-7.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of venetoclax combined with azacitidine regimen for newly diagnosed T-ALL patients.

DETAILED DESCRIPTION:
This is a phase 2, open Label, single arm, multi-center study for newly diagnosed T-cell acute lymphoblastic leukemia patients. The patients will receive vanetoclax combined with azacitidine as the induction regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 15.
2. Patients diagnosed with T-ALL according to 2016 WHO criteria for precursor lymphoid neoplasms.
3. ECOG performance status score less than 3.
4. Patients without serious heart, lung, liver, or kidney dysfunction.
5. Ability to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures.
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
3. Patients with uncontrolled active infection
4. Patients with active bleeding.
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
6. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met.
7. Liver dysfunction (total bilirubin > 1.5 times the upper limit of the normal range, ALT/AST > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value).
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
9. Surgery on the main organs within the past six weeks.
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results.
11. Patients who have received chemotherapy treatments related to the disease.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | At the end of Cycle 1 (each cycle is 21 days)
  The overall response (complete remission, complete remission with incomplete blood count recovery) rate achieved after one or two courses (21 days) induction therapy by venetoclax combined azacitidine regimen.

SECONDARY OUTCOMES:
Overall survial (OS) | 2 years
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Progression-Free Survival (PFS) | 2 years
  It is measured from the date of entry into this trial to the date of progression or death.
Number of adverse events | 2 years
  Adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No